CLINICAL TRIAL: NCT00140725
Title: A Randomised Trial of Lamivudine Plus Interferon Versus Lamivudine for the Treatment of HBeAg Positive Chronic Hepatitis B Virus (HBV)
Brief Title: Lamivudine Plus Interferon Versus Lamivudine For The Treatment Of HBeAg Positive Chronic Hepatitis B Virus (HBV)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Study Director, GSK
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NUC30938
Record Dates: First submitted 2005-08-31; First posted 2005-09-01 (Estimated); Last update posted 2008-10-16 (Estimated); Status verified 2008-10

CONDITIONS: Chronic Hepatitis B
Keywords: HBeAg-positive; chronic; Hepatitis B; lamivudine; seroconversion; Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic; Bronchiolitis Obliterans Syndrome; Hepatitis B; HIV Seropositivity | interventions — Lamivudine

INTERVENTIONS:
Drug: Lamivudine plus Polyethylene glyco-interferon alfa-2b
Drug: Lamivudine
  Other Names: Lamivudine plus Polyethylene glyco-interferon alfa-2b

SUMMARY:
This is a single-centre prospective randomised study comparing the virological and histological response of HBV infection to lamivudine in combination with interferon versus lamivudine alone.

ELIGIBILITY:
Inclusion criteria:

* Untreated chronic hepatitis B patients with evidence of HBV replication as documented by serum HNV-DNA positive within 3 months prior to entry and serum HBeAg positive at screening.
* Documented presence of abnormal alanine aminotransferase (ALT) (1.3 - 5X upper limit normal (ULN)) within 1 month prior to entry and signs of compensated liver disease.

Exclusion criteria:

* Patients with any cause for liver disease other than chronic hepatitis B and evidence or history of decompensated liver disease.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160
Dates: Start 2000-04

PRIMARY OUTCOMES:
Proportion of patients with HBeAg seroconversion to anti-HBe

SECONDARY OUTCOMES:
Normalization of alanine aminotransferase (ALT)
Undetectable HBV DNA
Histologic improvement
Tyrosine, methionine, aspartate, aspartate (YMDD) mutants among the viremic relapsers at the end of therapy and safety of treatment

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, MD, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Shatin, Hong Kong